CLINICAL TRIAL: NCT05029947
Title: Setting Benchmarks for Microsurgical Clipping of Unruptured Intracranial Aneurysms - An Analysis of Standardized Outcome References From an International Multicentre Cohort
Brief Title: Setting Benchmarks for Microsurgical Clipping of Unruptured Intracranial Aneurysms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Richard Drexler, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: BenchmarkUIA
Record Dates: First submitted 2021-08-29; First posted 2021-09-01 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Aneurysm; Aneurysm, Brain; Aneurysm Cerebral; Aneurysm of Cerebral Artery; Aneurysm, Intracranial
MeSH Terms: conditions — Aneurysm; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Microsurgical Clipping of Unruptured Intracranial Aneurysm — Microsurgical Clipping of Unruptured Intracranial Aneurysm

SUMMARY:
To conduct a retrospective multicenter cohort study to define benchmark values for best achievable outcomes following microsurgical clipping of unruptured intracranial aneurysms (UIA).

DETAILED DESCRIPTION:
Surgeons strive for the best possible outcome of their surgeries with the greatest possible chance for recovery of the patients. Therefore, monitoring and quality improvement is increasingly important in surgery. For this purpose, different concepts were developed with the aim to assess best achievable results for several surgical procedures and reduce unwarranted variation between different centers. The concept of a benchmark establishes reference values which represents the best possible outcome of high-volume centers and can be used for comparison and improvement. In the past years, the concept of benchmarking attaches greater importance in the field of healthcare, especially in surgery. Benchmark values are established within a patients' cohort for which the best possible outcome can be expected. The aim of our study is the establishment of robust and standardized outcome references after microsurgical clipping of unruptured intracranial aneurysms. After successful implementation of benchmarks from an international cohort of renowned centers, these data serve as reference values for the evaluation of novel surgical techniques and comparisons among centers or future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients who went through elective microsurgical clipping of unruptured intracranial aneurysm
* High-volume centers with ≥40 cases per year during the study period

Exclusion Criteria:

* Treatment following subarachnoid haemorrhage
* Clipping following an incomplete occlusion after previous treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who went through elective microsurgical clipping of unruptured intracranial aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete occlusion of aneurysm | up to 6 months
  Aneurysm remnant in CT scan or angiography
Retreatment of aneurysm | up to 6 months
  Necessity of retreatment in endovascular or microsurgical technique
Mortality | up to 6 months
  Death of the patient

SECONDARY OUTCOMES:
Chronic subdural hematoma | up to 6 months
  Development of chronic subdural hepatoma requiring intervention
Stroke | up to 6 months
  Occurrence of ischemic stroke
Cerebral vasospasm | up to 6 months
  Occurrence of cerebral vasospasm
Intracerebal haemorrhage | up to 6 months
  Occurrence of intracerebral haemorrhage related to aneurysm treatment
New neurological deficit | up to 6 months
  None, motor deficit, sensory deficit, aphasie
Modified Rankin Score | up to 6 months
  Difference of mRS compared to preoperative status
Glasgow Outcome Scale | up to 6 months
  From 1 (death) to 5 (low disability)

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Dührsen, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany